CLINICAL TRIAL: NCT00065780
Title: Ventricular Size and Value Calcification Measures by Computed Tomography - Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Other Study IDs: 1231; R01HL071739 (NIH)
Record Dates: First submitted 2003-07-31; First posted 2003-08-04 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To rescan 6,700 subjects in the MESA study to obtain computed tomography measures of calcification.

DETAILED DESCRIPTION:
BACKGROUND:

This study is ancillary to the MultiEthnic Study of Atherosclerosis (MESA) Trial, a prospective investigation of the etiology and natural history of atherosclerosis and the ability of non-invasive tools to measure atherosclerotic burden and identify high risk individuals in a large, population-based cohort. The development of computed tomography (CT) to evaluate coronary calcification (CC) now provides a tool to directly measure coronary atherosclerosis non-invasively. The information obtained by CT however provides more information than CC alone. CT has the ability to measure and quantitate aortic valve calcification (AVC), mitral annular calcification (MAC), aortic wall calcification and left ventricular size (LVS). The longitudinal nature of this study will allow epidemiologic associations to be established for a multitude of risk factors and these measures, establishing both the time sequence for each measure and consistency of the association in a variety of populations (ethnicity, gender, geographical location and age). Magnetic resonance imaging of the heart will also be obtained as part of the MESA trial, and comparisons of LV size by CT to magnetic resonance measures will also be performed.

DESIGN NARRATIVE:

This study is ancillary to the MultiEthnic Study of Atherosclerosis (MESA) Trial, a prospective investigation of the etiology and natural history of atherosclerosis and the ability of non-invasive tools to measure atherosclerotic burden and identify high risk individuals in a large, population-based cohort. The development of computed tomography (CT) to evaluate coronary calcification (CC) now provides a tool to directly measure coronary atherosclerosis non-invasively. The information obtained by CT however provides more information than CC alone. CT has the ability to measure and quantitate aortic valve calcification (AVC), mitral annular calcification (MAC), aortic wall calcification and left ventricular size (LVS). The longitudinal nature of this study will allow epidemiologic associations to be established for a multitude of risk factors and these measures, establishing both the time sequence for each measure and consistency of the association in a variety of populations (ethnicity, gender, geographical location and age). Magnetic resonance imaging of the heart will also be obtained as part of the MESA trial, and comparisons of LV size by CT to magnetic resonance measures will also be performed. The investigators will utilize scans already obtained as part of the calcium scanning (at baseline and 3.5 year follow-up), and make these four measures on baseline and follow-up scans obtained. The additive value of these simple measures to CC score could possibly provide clinicians with even more power to identify and stratify the high-risk cardiac patient with both findings. This study will also establish the prevalence, in a population based study, of all both AVC and MAC, using a technique highly sensitive to see these abnormalities. It has been postulated that a 'total atherosclerotic burden' could be obtained by adding CAC to thoracic aortic calcification, and this total atherosclerosis score (with or without MAC and AVC) might better predict cardiovascular events than CAC alone. Similarly, this cohort of 6,700 patients with repeat scans can be assessed for factors that enhance or inhibit progression of LVS, mitral annular, aortic valve or wall calcification, lending insight into therapies that have efficacy against progression of aortic sclerosis or left ventricular enlargement.

ELIGIBILITY:
No eligibility criteria

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MESA study population - 6814 participants from 6 clinic sites around the US
Sampling Method: Probability Sample
Enrollment: 6814 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Valve Calcification | 2002, again in 2004-5
  valve calcification of aortic and mitral valve
Aortic valve calcification | 2002, again in 2004-2005
  valve calcification of the aortic valve on cardiac ct